CLINICAL TRIAL: NCT05064306
Title: Expanded Access Use of 131I-Omburtamab Intraventricular Radioimmunotherapy for Central Nervous System/Leptomeningeal Neoplasms
Brief Title: 131I-omburtamab for the Treatment of Central Nervous System/Leptomeningeal Neoplasms in Children and Young Adults
Status: No longer available | Type: Expanded Access
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-345
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Central Nervous System/Leptomeningeal Neoplasms
Keywords: 131I-omburtamab; neuroblastoma; medulloblastoma; rhabdoid tumors; pineoblastoma; retinoblastoma; PNET; rhabdomyosarcoma; Ewing's sarcoma; Wilm's tumor; hepatoblastoma; non-embryonal tumors; histologic confirmation of B7-H3 reactivity; 21-345
MeSH Terms: conditions — Meningeal Neoplasms; Neuroblastoma; Medulloblastoma; Rhabdoid Tumor; Pinealoma; Retinoblastoma; Neuroectodermal Tumors, Primitive; Rhabdomyosarcoma; Sarcoma, Ewing; Wilms Tumor; Hepatoblastoma | interventions — omburtamab I-131

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: 131I-omburtamab — 50 mCi 131I-omburtamab

SUMMARY:
The researchers are doing this study to provide access to treatment with 131I-omburtamab for children and young adults who have CNS/leptomeningeal neoplasms. 131I-omburtamab is an investigational drug; the FDA has not approved it to treat this cancer or any other disease. However, the agency has granted the drug Breakthrough Therapy Designation for the treatment of neuroblastoma with CNS metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of an embryonal malignancy (including but not limited to neuroblastoma, medulloblastoma, rhabdoid tumors, pineoblastoma, retinoblastoma, PNET, rhabdomyosarcoma, Ewing's sarcoma, Wilm's tumor, hepatoblastoma) other non-embryonal tumors must have histologic confirmation of B7-H3 reactivity.
* Patients must have a diagnosis of CNS/ leptomeningeal disease which has been treated with conventional therapies or for which no conventional therapy exists or a recurrent brain tumor with a predilection for leptomeningeal dissemination (i.e. PNET, rhabdoid tumor).
* Chemotherapy:

  °Patients must have received their last dose of myelosuppressive anticancer therapy at least 21 days (3 weeks) prior to receiving treatment dose(s).
* Biologic or investigational agent (anti-neoplastic):

  * Patients who are currently on biological (small molecule inhibitors such as ALK inhibitors, ROS inhibitors or MEK inhibitors etc.) or investigational agents that are considered non-myelosuppressive can continue treatment but should have recovered from any acute toxicity potentially related to the agent.
  * Patients may be treated if they received one prior treatment dose with 131I-omburtamab
* Monoclonal antibody treatment and agents with known prolonged half-lives:

  * Patients must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 21 days prior to enrollment.
  * Monoclonal antibody treatment and agents with known prolonged half-lives: Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the agent ≥ 28 days prior to receiving treatment dose(s).
* Neurologic Status:

  * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment.
  * Patients with seizure disorders may be enrolled if seizures are controlled.
* Performance Status:

  °Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within 2 weeks prior to study enrollment must be ≥ 50%. Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate bone marrow function defined as:

  * Peripheral absolute neutrophil count (ANC) ≥ 0.5x 10^9/ L (must not have received G-CSF within the 7 days prior to enrollment or pegfilgrastim within the 14 days prior to enrollment)
  * Platelet count ≥ 50 x 10^9/ L (unsupported, defined as no platelet transfusion within 7 days prior to study enrollment)
* Intraventricular Access Device °Protocol treatment with radioimmunotherapy (131I-omburtumab) will require the presence of an appropriate intraventricular access device (e.g.,programmable ventriculoperitoneal [VP] shunt or Ommaya reservoir). Patients are not required to have an existing programmable VP shunt or Ommaya at the time of study enrollment but must be willing and able to undergo a surgical procedure to have one placed prior to Radioimmunotherapy.

Note: Patients with an existing intraventricular VP shunt without a programmable component must be willing and able to undergo modification of the shunt before treatment with 131I-omburtumab.

* Both pediatric and adult patients of any age are eligible.
* Patients may have active malignancy outside the central nervous system.
* Patients may be on standing steroids, as long as the dosage is either stable or decreasing for at least week prior to enrollment
* Signed informed consent and assent when appropriate indicating awareness of the investigational nature of this study.

Exclusion Criteria:

* Patients with obstructive or symptomatic communicating hydrocephalus
* Patients with an uncontrolled life-threatening infection
* Patients who are pregnant: negative pregnancy test is required for all women of childbearing age, and appropriate contraception is required during the study period.
* Patients who have received cranial or spinal irradiation less than 3 weeks prior to first dose

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Farouk Sait, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm